CLINICAL TRIAL: NCT03723291
Title: PentoxIfylline and Tocopherol for the Treatment of Post-radiotherapy Fibrosis in Head and Neck Cancer Patients: a Feasibility Study
Brief Title: PentoxIfylline and Tocopherol for the Treatment of Post-radiotherapy Fibrosis in Head and Neck Cancer Patients
Acronym: PITSTOP
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15/0483
Record Dates: First submitted 2018-10-24; First posted 2018-10-29 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Head and Neck Fibrosis
Keywords: Head and Neck
MeSH Terms: interventions — alpha-Tocopherol; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Intervention Model Description: Multicentre, parallel group, randomised controlled trial in 50 patients with radiotherapy-induced fibrosis of the head and neck.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): The current best standard of care [rehabilitation exercises]
  Interventions: Procedure: • Arm A: Best standard of care only [a structured programme of rehabilitation exercises] for 6 months
- Arm B (Experimental): The current best standard of care [rehabilitation exercises] + the experimental intervention
  Interventions: Combination Product: Arm B: A combination of pentoxifylline and tocopherol acetate in addition to best standard care [a structured programme of rehabilitation exercises] for 6 months

INTERVENTIONS:
Combination Product: Arm B: A combination of pentoxifylline and tocopherol acetate in addition to best standard care [a structured programme of rehabilitation exercises] for 6 months — • Arm B: A combination of pentoxifylline 800 mg/d in two 400-mg tablets and 1,000 IU/d of tocopherol acetate in two 500-IU aliquots in addition to best standard care [a structured programme of rehabilitation exercises] for 6 months
  Arms: Arm B
Procedure: • Arm A: Best standard of care only [a structured programme of rehabilitation exercises] for 6 months — Prophylactic swallowing exercises consist of strap muscle exercises, airway protection exercises and base of tongue exercises
  Arms: Arm A

SUMMARY:
Objectives:

This is a feasibility study in preparation for the main multicentre randomised trial, which is anticipated to have two arms:

* Arm A: the current best standard of care [rehabilitation exercises]
* Arm B: the current best standard of care [rehabilitation exercises] + the experimental intervention

In this feasibility trial the following aspects will be evaluated:

* Recruitment rates [that is also willingness to be randomised]
* Feasibility of providing the experimental intervention at the NHS study sites
* Retention rate/drop out rate
* Feasibility and acceptability of (i) proposed primary outcome [patient-centred], (ii) a range of additional patient-centred and clinician-centred outcomes
* Standard deviation of the proposed primary outcome so to inform sample size calculation of the main trial.
* Safety/toxicity of the study medication.

Type of trial: Multicentre, parallel group, randomised controlled trial in 50 patients with radiotherapy-induced fibrosis of the head and neck.

Trial design and methods:

Participants over the age of 18, with radiotherapy-induced fibrosis of the head and neck will be given information about the trial and invited to participate.

50 participants who consent will be recruited and randomised to either:

* Treatment with pentoxifylline 400 mg tablets twice a day [total 800mg/day] + 500IU tocopherol acetate solution twice a day [total 1000 IU/day] in addition to best standard care [a structured programme of rehabilitation exercises] for 6 months or
* Best standard of care [a structured programme of rehabilitation exercises] for 6 months.

Randomisation will be carried out online

Trial duration per subject: 6 months Estimated total trial duration: 56 months Planned trial sites: Multi-site Total number of subjects planned: 50 participants

Main inclusion/exclusion criteria:

Inclusion Criteria:

* Subjects aged ≥18 years
* Previous history of Head & Neck Cancer
* Previous radiotherapy to the Head & Neck - minimum 50 Gy completed at least 12 months before screening visit
* Cancer-free for a minimum of 12 months after completion of radiotherapy.
* Diagnosis of radiotherapy-induced fibrosis of the head and neck: trismus and/or dysphagia

Exclusion Criteria:

* History of primary cancer resection and/or reconstructive surgery to anatomical areas involved in swallowing and/or chewing.
* Concomitant presence of other disorders that may cause pharyngeal/oral fibrosis
* Known hypersensitivity to pentoxifylline or tocopherol (vitamin E).
* History of acute porphyrias or haemorrhagic disorders
* Active/ongoing hypotension
* Diabetes
* Pregnancy
* Subjects with osteoradionecrosis
* Breastfeeding mothers
* Subjects with a MIO <12mm

Statistical methodology and analysis: Analysis of this feasibility trial will be mainly descriptive, measuring recruitment rate, acceptance of randomisation, attrition from treatment and trial, and completion rates for the outcome measures (to gauge acceptability and appropriateness).

DETAILED DESCRIPTION:
Fibrosis is a common and irreversible adverse effect of radiotherapy. Radiotherapy is used with curative intent in most individuals (~70%) with head and neck cancer (HNC), often in combination with surgery and/or chemotherapy. It is estimated that up to 60% of these individuals will experience persistent fibrosis as a toxic effect of the radiotherapy including trismus and dysphagia. As 680,000 new HNC cases/year are diagnosed worldwide, it is estimated that approximately 270,000 individuals will develop persistent trismus and/or dysphagia, with consequent reduced quality of life (QoL) due to impaired talking, eating, chewing and swallowing. Malnutrition, psychological and social issues add further suffering to affected individuals. Mortality is also significantly increased due to aspiration pneumonia. In the UK there are ~10,000 new H&N cancer cases/year, which translates into approximately 4,200 individuals experiencing radiotherapy-induced fibrosis (RIF) every year. Increasing incidence rates of H&N cancer suggest that these figures will increase over the next few years. This group of cancer survivors represent a challenge for the NHS: they have a chronic condition reducing their quality of life and no realistic therapeutic option as no intervention has proven long-term effective. Current best NHS practice consists of rehabilitation therapy (exercises). Although available literature suggests potential efficacy, evidence is very weak: relevant benefits seem to be short-lived, the effect size is usually small, and compliance with treatment is often poor. As preparatory work for this proposal we have performed a systematic review of the literature, which shows that five prospective studies investigated rehabilitation exercises, pentoxifylline and botulinum A in the therapy of post-RT trismus. Four prospective studies investigated rehabilitation exercises and electrical stimulation in the therapy of post-RT dysphagia.

Overall studies were at high risk of bias, and there was very limited evidence supporting the efficacy of the above interventions in the post-RT setting.

There remains little ongoing clinical research in this field at the present moment (clinical trials databases searched in March 2018). Most ongoing recruiting studies focus on preventive strategies during HNC radiotherapy. In terms of trials aimed at reducing established post-RT fibrosis, we could only find one recruiting Canadian study on manual therapy and one American study on self-care program, with no UK study.

RIF has been traditionally considered an irreversible disorder characterised by the generation of reactive oxygen species, vascular damage, pro-fibrotic inflammation, promotion of collagen formation and the development of excessive fibrous tissue. However research during the last 15 years has shown that co-administration of pentoxifylline and tocopherol (vitamin E) can reduce and reverse the fibrotic process. Pentoxifylline is known to improve microcirculation, inhibit fibroblast proliferation, reduce extracellular matrix production, and increase collagenase activity. Tocopherol (Vitamin E) has antioxidant properties. The precise mechanisms by which the pentoxifylline/tocopherol (vitamin E) combination interacts with fibro-atrophic tissues and induces fibrotic process reversibility are still unclear. It has been suggested that the anti-fibrotic effects are consequence of the inhibition of fibroblast proliferation and extracellular matrix production, increased collagenase activity, as well as a reduction in reactive oxygen species. Clinical trials have indicated that the combination of pentoxifylline and tocopherol (vitamin E) can decrease and even reverse RIF in individuals irradiated to the breast, pelvis, lung, and prostate, leading to functional and aesthetic benefits. It is not known whether this therapy may have similar beneficial effects in HNC survivors with permanent RIF (trismus and/or dysphagia). Preliminary small-scale studies suggest that this may be the case, and support the notion that pentoxifylline and tocopherol (vitamin E) represent a promising treatment that is worth investigating in well-designed clinical trials. The best available evidence comes from a 2001 uncontrolled, small (16 subjects) pilot study that showed functional improvement in subjects with established post-radiotherapy trismus after an 8-week course of pentoxifylline as monotherapy. Other studies have reported the beneficial effects of pentoxyfilline monotherapy or in combination with tocopherol (vitamin E) in reducing and/or preventing RIF in HNC, but these focused on cutaneous/subcutaneous neck fibrosis and did not measure trismus/dysphagia. There is a clear need for better-designed clinical research as more robust evidence is required in order to influence changes in NHS practice and improve the quality of life of HNC survivors.

The main study will be a multicentre randomised controlled trial with two arms including the experimental intervention plus the current best standard treatment versus the current best treatment as comparator [1:1]. The main outcome will be anticipated to be patient-centred and measured via a validated instrument (QoL questionnaire), with secondary outcomes including other patient-centred measures (validated functional questionnaires) as well as clinician-rated and instrumental outcomes. However several aspects of the main trial remain unknown/unclear and would require clarification via a feasibility study.

PITSTOP is a feasibility 36-month randomised trial of the best standard therapy alone [rehabilitation exercises] vs treatment with pentoxifylline and tocopherol (vitamin E) in addition to best standard therapy (rehabilitation exercises) in 50 participants with radiotherapy-induced fibrosis of the head and neck. It is a two-centre study with a 1:1 randomisation into two study arms. At each site a blocked randomisation list will be used to ensure an approximate balance in numbers between the two groups. Allocation concealment will be ensured using an online randomisation service (Sealed Envelope).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged ≥18 years at the time of signing the Informed Consent Form
* Subjects with diagnosis of radiotherapy-induced fibrosis of the head and neck: trismus and/or dysphagia as defined by the following patient-centred criteria: Trismus: "Does your mouth opening feel restricted" (answer must be yes). Dysphagia: a score of 3 or more on the 10-item Eating Assessment Tool (EAT-10)
* Previous History of Head & Neck Cancer
* Previous radiotherapy to the Head & Neck - minimum 50 Gy completed at least 12 months before screening visit
* No history of primary cancer resection and/or reconstructive surgery to anatomical areas involved in swallowing and/or chewing with potential for altered and reconstructed muscular anatomy that may not be amenable to exercise/respond to anti-fibrotic medications (with the exception of diagnostic biopsy/tonsillectomy and neck lymphadenectomy)
* Cancer-free for a minimum of 12 months after completion of radiotherapy, (complete clinical/radiological remission; absence of distant metastases)
* Able to understand the purpose of the study and willing to sign informed consent.
* Able to take study medications orally
* Subjects of child bearing potential/potency must adhere to one method of highly effective contraception.
* Subject has provided written informed consent

Exclusion Criteria:

* Concomitant presence of other disorders that may cause trismus or dysphagia (e.g. active temporomandibular joint disorder limiting mouth opening, scleroderma, oral sub mucous fibrosis or other rheumatological or neurological disease)
* Subject has recurrent H&N cancer or second primary H&N cancer
* Subject has a known hypersensitivity to pentoxifylline or other xanthines such as caffeine, theophylline and theobromine or tocopherol (vitamin E).
* Subject has a history of acute porphyrias (acute intermittent porphyria, variegate porphyria, hereditary coproporphyria and 5-aminolaevulinic acid dehydratase deficiency porphyria)
* Subject has a history of cerebral haemorrhage, extensive retinal haemorrhage or is at risk of increased bleeding including those taking anticoagulants and platelet aggregation inhibitors such as: clopidogrel, eptifibatide, tirofiban, epoprostenol, iloprost, abciximab, anagrelide, NSAIDs other than selective COX-2 inhibitors, acetylsalicylates (ASA/LAS), ticlopidine, dipyridamole
* Subject has a history of acute myocardial infarction, coronary artery disease, cardiac arrhythmias
* Subject has a active/ongoing hypotension*
* Subject has a active/ongoing hepatic or renal impairment*
* Subject has a history of diabetes*
* Expected non-compliance with treatment interventions or is considered unsuitable for trial participation at the discretion of the treating clinician.
* Current pregnancy as confirmed by urine pregnancy test at screening.
* Patients with rare hereditary problems of fructose intolerance, glucose-galactose malabsorption or sucrase-isomaltase insufficiency.
* Subjects with osteoradionecrosis of the jaw.
* Breastfeeding mothers
* Subjects with a MIO of <12mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate achieved | 36 months
  Proportion of eligible subjects who consent to be randomised
Usable EORTC H&N35 scores | 6 months
  Proportion of randomised subjects who have a useable (non missing) score for the EORTC QLQ-H&N35 questionnaire at 6 months (this is a validated H&N Radiotherapy-specific QoL questionnaire for both trismus and dysphagia which we expect to provide the primary outcome for the main trial). Thsi scale runs from 1-4 with 4 being very much and 1 not at all.

SECONDARY OUTCOMES:
Proportion of drop out over 6 months | 6 months
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability of Pentoxifylline & Tocopherol] | 36 months
  The safety of Pentoxifylline and Tocopherol will be assessed through adverse event recording
Proportion of randomised subjects who have useable (non missing) scores for Validated QoL questionnaire for Dysphagia: the M.D. Anderson Dysphagia Inventory (MDADI) | 6 months
Proportion of randomised subjects who have useable (non missing) scores for Validated functional questionnaire for Dysphagia: 10-item Eating Assessment Tool (EAT-10) | 6 months
Proportion of randomised subjects who have useable (non missing) scores for Validated functional questionnaire for Trismus: the Gothenburg Trismus Questionnaire | 6 months
Proportion of randomised subjects who have useable (non missing) scores for Validated Oral Health-related QoL questionnaire: EORTC QLQ-OH15 | 6 months
Proportion of randomised subjects who have useable (non missing) scores for Validated European Organisation for Research and Treatment of Cancer Core Questionnaire - Quality of Life of Cancer Patients (EORTC QlQ-C30) | 6 months
Proportion of randomised subjects who have useable (non missing) scores for Clinical Global Impression Scales for Trismus: a 5-point scales will be used to allow subjects to rate perceived post-treatment changes in their trismus | 6 months
Proportion of randomised subjects who have useable (non missing) scores for Clinical Global Impression Scales for Dysphagia: a 5-point scales will be used to allow subjects to rate perceived post-treatment changes in their dysphagia | 6 months
Proportion of randomised subjects who have useable (non missing) scores for National Cancer Institute Common Terminology Criteria for Adverse Events scale (NCI-CTCAEv4) -grading for Trismus | 6 months
Proportion of randomised subjects who have useable (non missing) scores for NCI-CTCAEv4 - grading for Dysphagia | 6 months
Proportion of randomised subjects who have useable (non missing) scores for Trismus: Measurement of mouth opening (recorded using Willis bite calliper) | 6 months
Proportion of randomised subjects who have useable (non missing) scores for Dysphagia: Videofluoroscopy [VFS] with Penetration Aspiration Scale, DIGEST grade and 100ml Water Swallow Test (Volume, Capacity and Speed scores) | 6 months
Proportion of randomised subjects who have useable (non missing) scores for PSS-HN - performance scales rated by health professionals, normalcy of diet, public eating and understandability of speech | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Aintree University Hospital NHS Foundation Trust, Liverpool
  - University College London Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No